CLINICAL TRIAL: NCT05911152
Title: Safety and Feasibility of Laparoscopic Intracorporeal Anastomosis for Colorectal Surgery- A Multiple Center Real World Study
Acronym: SELECTED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC4050
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Minimally invasive surgery; Laparoscopic surgery; Intracorporeal anastomosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracorporeal anastomosis: Patients underwent laparoscopic colorectal surgery with intracorporeal anastomosis
  Interventions: Procedure: Intracorporeal anastomosis
- Extracorporeal anastomosis: Patients underwent laparoscopic colorectal surgery with extracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — Surgeons perform totally laparoscopic intracorporeal digestive reconstruction after specimen resection
  Groups: Intracorporeal anastomosis

SUMMARY:
The goal of this observational study is to explore the safety and feasibility of laparoscopic intracorporeal anastomosis in colorectal cancer surgery. The main questions it aims to answer are: 1. If intracorporeal anastomosis is safe in terms of short-term outcome? 2. If intracorporeal anastomosis can achieve the same oncological outcome as conventional extracorporeal anastomosis?

DETAILED DESCRIPTION:
This study is a retrospective real-world research initiated by the Chinese Academy of Medical Sciences Cancer Hospital, including Cancer Hospital of the Chinese Academy of Medical Sciences, Shenzhen Hospital and Peking University First Hospital. The study aims to retrospectively analyze the clinical data of approximately 2,000 patients who underwent laparoscopic surgery with preoperative imaging staging of cT1-4aNanyM0 and pathological diagnosis of adenocarcinoma or high-grade intraepithelial neoplasia from April 2016 to April 2020. The patients will be divided into the intracorporeal anastomosis group (IA) and extracorporeal anastomosis group (EA) based on the surgical records. The primary endpoints of the study are 3-year disease-free survival (DFS) and 3-year overall survival (OS). The secondary endpoints include overall complication rate within 30 days, postoperative pain score, time to first flatus after surgery, time to first bowel movement after surgery, time to first oral intake after surgery, length of hospital stay, and postoperative quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily enrolled in this study and signed an informed consent form;
2. Age: 18-75 years;
3. Completion of colonoscopy and biopsy, with pathological confirmation of adenocarcinoma or high-grade intraepithelial neoplasia;
4. Preoperative enhanced CT or MRI examination showing no evidence of distant metastasis;
5. Preoperative staging as cT1-3NanyM0;
6. Underwent laparoscopic surgery.

Exclusion Criteria:

1. Contraindications to laparoscopic surgery;
2. Cases requiring emergency surgery due to acute bowel obstruction, perforation, or bleeding;
3. Patients with distant metastasis;
4. Patients with multiple primary colorectal cancers;
5. Patients with a history of malignancy;
6. Patients unwilling to sign the informed consent or unwilling to follow the study protocol for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent laparoscopic colorectal surgery with intracorporeal or extracorporeal anastomosis
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 year
  Proportion of patients who remain alive without any signs or symptoms of disease recurrence or progression for a period of 3 years after surgery
3-year overall survival | 3 year
  Percentage of patients who are still alive at the end of a 3-year period after surgery

SECONDARY OUTCOMES:
Rate of postoperative complications | 30 days
  Rate of postoperative complications within 30 days after surgery
Time to first flatus after surgery | 7 days
  Time to first flatus after surgery
Time to first stool after surgery | 7 days
  Time to first stool after surgery
Length of stay after surgery | 30 days
  Length of stay after surgery
Postoperative pain score | 3 days
  VAS (Visual Analog Scale) score is used to assess the postoperative pain level in patients. It is a measurement tool used to assess the intensity or severity of a subjective experience, typically related to pain or discomfort. The VAS score involves a straight line or a numerical scale ranging from 0 to 10, where 0 represents no pain or discomfort and 10 represents the worst possible pain or discomfort. Individuals are asked to indicate their level of pain or discomfort by marking a point on the scale, and the score is determined by measuring the distance from the 0 mark to the marked point. The VAS score provides a subjective assessment of pain or discomfort experienced by an individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang M, Dong S, Wang L, Liu Z, Zhou H, Liu Q, Chen Y, Tang J, Wang X. Short-term and long-term outcomes of intracorporeal anastomosis in laparoscopic segmental left colectomy for splenic flexure cancer - a multicenter retrospective cohort study of 342 cases. Int J Surg. 2024 Mar 1;110(3):1595-1604. doi: 10.1097/JS9.0000000000000974. PMID 38085798